CLINICAL TRIAL: NCT05526885
Title: Tuberculosis Diagnostic Trial of CAD4TB Screening Alone Compared to CAD4TB Screening Combined With a CRP Triage Test, Both Followed by Confirmatory Xpert MTB/RIF Ultra in Communities of Lesotho and South Africa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klaus Reither (Other)
Collaborators: SolidarMed (Other); Institute of Tropical Medicine, Belgium (Other); Radboud University Medical Center (Other); Charite University, Berlin, Germany (Other); Human Sciences Research Council (Other Government)
Responsible Party: Sponsor-Investigator, Klaus Reither, Head of Clinical Research Unit, Swiss Tropical & Public Health Institute
Organization: Swiss Tropical & Public Health Institute (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P1685-22B
Record Dates: First submitted 2022-08-31; First posted 2022-09-02 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Tuberculosis
Keywords: Lesotho; South Africa; community-based; tuberculosis; active case findings; cost-effectiveness; CAD4TB; POC-CRP; Xpert MTB/RIF Ultra; triage; screening
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Intervention Model Description: In this study a paired screen-positive design is used to directly compare two screening/triage approaches in the same individual based on a paired analysis: CAD4TB screening only (approach 1) versus CAD4TB screening with POC-CRP triage algorithm (approach 2).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Approach 1 - CAD4TB screening (Experimental): Participants with a CAD4TB version 7 (Delft Imaging, NL) score above the overall threshold (as defined for study approach 1) are eligible for Xpert MTB/RIF Ultra testing.
  Interventions: Diagnostic Test: CAD4TB; Diagnostic Test: Xpert MTB/RIF Ultra
- Approach 2 - CAD4TB screening with POC-CRP triage testing (Experimental): Participants with a CAD4TB version 7 (Delft Imaging, NL) score within the threshold window (between lower and upper limit threshold as defined for study approach 2), a POC-CRP LumiraDx (LumiraDx Limited, UK) test will follow as a triage test. If CRP is above the determined threshold as defined for approach 2, Xpert MTB/RIF Ultra will be performed. If the CAD4TB score is above the upper limit threshold as defined for approach 2, Xpert MTB/RIF Ultra will be performed (without further CRP testing).
  Interventions: Diagnostic Test: CAD4TB; Diagnostic Test: POC-CRP; Diagnostic Test: Xpert MTB/RIF Ultra

INTERVENTIONS:
Diagnostic Test: CAD4TB — A posterior anterior digital chest X-ray incoporated in a mobile diagnostic unit is analysed by CAD4TB version 7 (Delft Imaging, NL). A trained and qualified person in compliance with national regulations will operate the digital chest X-ray.
Diagnostic Test: POC-CRP — A quantitative POC-CRP LumiraDx (LumiraDx Limited, UK) triage test will be performed by finger-prick if CAD4TB scores is within the defined threshold window of study approach 2 triage testing
  Arms: Approach 2 - CAD4TB screening with POC-CRP triage testing
Diagnostic Test: Xpert MTB/RIF Ultra — Depending on CAD4TB (approach 1 & 2) or POC-CRP score (approach 2) a confirmatory Xpert MTB/RIF Ultra(Cepheid, USA) rapid sputum molecular testing follows for both Mycobacterium tuberculosis complex and rifampicin resistance;

SUMMARY:
According to WHO, about 40% of the incident TB cases in 2020 are either under-reported or under-diagnosed causing on one hand major health risks and on the other hand catastrophic financial consequences. In particular, indigent people in hard-to-reach communities with high TB/HIV burden are at high risk of missed or delayed diagnoses. Hence, active case finding for TB remains an integral part of tuberculosis control in high-risk groups, such as people living with HIV (PLHIV) or diabetes mellitus, people living in specific geographical locations associated with a high burden of TB and poor access to health care, miners, or prisoners. CAD4TB (Delft Imaging, NL), a digital chest X-ray analysis software, and point-of care C-reactive protein assay (POC-CRP; e.g. LumiraDx, UK), which detects a cytokine induced acute phase protein, are two tests which have great potential of becoming a screening and triage test for TB as outlined in the WHO target product profiles. Data on CAD4TB and CRP suggest that accuracy can be improved if thresholds are stratified by patient characteristics, such as HIV status, history of TB and TB symptoms. TB TRIAGE+ Trial takes place in the communities of Lesotho and South Africa, which present high prevalence of subclinical TB, where a symptom-based screening would miss almost half of all infectious TB cases. TB TRIAGE+ Trials conducts a direct (in the same individual) comparison of the two screening/triaging approaches which are not based on symptoms: CAD4TB screening alone (approach 1) versus CAD4TB screening with POC-CRP triage testing (approach 2), and followed by confirmatory Xpert MTB/RIF Ultra testing in both approaches. TB TRIAGE TRIAL is investigates the hypothesis that a community-based active case finding strategy with CAD4TB screening with POC-CRP triage testing (approach 2) will be non-inferior compared to CAD4TB screening alone (approach 1) with regard to yield of detected TB cases and superior with regard to cost effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide signed written consent or witnessed oral consent in the case of illiteracy, prior to undertaking any study-related procedure
* Adults (≥18 years)

Exclusion Criteria:

* Any condition for which participation in the study, as judged by the investigator or a designated staff member, could compromise the well-being of the subject or prevent, limit or confound protocol specified assessments
* Seriously ill person who needs immediate medical care
* Current anti-TB treatment (preventive TB treatment permitted)
* Lesotho only: Pregnancy (self-reported)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20000 (Actual)
Dates: Start 2022-09-07 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Yield of detected TB cases per study approach: number of positive Xpert MTB/RIF Ultra results per screening approach. | 24 Months
Cost-effectiveness of the CAD4TBv7-CRP approach using the CAD4TBv7 approach as a comparator: the costs for each positive Xpert Ultra case detected in the CAD4TBv7-CRP approach compared to the CAD4TBv7 approach | 24 Months

SECONDARY OUTCOMES:
Extension of primary outcome: Cost-effectiveness of the CAD4TBv7-CRP approach and the CAD4TBv7 approach compared to passive case finding: cost per TB case detected | 24 Months
Equity analysis: 1. Socioeconomic status of households with actively detected TB cases compared to those with passively detected TB cases and to households with no TB cases: wealth quintiles distribution, income distribution and main source of income | 24 Months
Equity analysis: 2. Average out of pocket payments (OOP) associated with accessing TB treatment for households with identified TB cases across different wealth quintiles | 24 months
Health impact: The expected number of identified TB cases via passive case finding if the active case finding campaign had not taken place will be compared to the number of cases identified in the campaign | 24 months

CONTACTS AND LOCATIONS:
Locations (2):
- SolidarMed, Maseru, Lesotho
- Human Sciences Research Council, Pietermaritzburg, KwaZulu-Natal, South Africa

IPD SHARING:
Plan to Share IPD: Yes
All data will be stored securely in a way that allows future access for the research team. We will adhere to the FAIR Guiding Principles for data management and stewardship. After completion of the studies and after anonymization (e.g. replace subject identifier with a new random subject identifier), analysis datasets will be made publicly available in a timely manner on a non-commercial data platform according to the FAIR principles.

REFERENCES:
- [Result] Signorell A, van Heerden A, Ayakaka I, Jacobs BK, Antillon M, Tediosi F, Verjans A, Brugger C, Harkare HV, Labhardt ND, Bosman S, Kamele M, Keitseng M, Madonsela T, Kurscheid J, Muhairwe J, Keter AK, Murphy K, van Ginneken B, Gils T, Katende B, Gebresenbet RF, Erhardt RM, Zoller T, Vanobberghen F, Glass TR, Lynen L, Reither K. Effectiveness and cost-effectiveness of community-based TB screening algorithms using computer-aided detection (CAD) technology alone compared with CAD combined with point-of-care C reactive protein testing in Lesotho and South Africa: protocol for a paired screen-positive trial. BMJ Open. 2025 Jul 28;15(7):e093989. doi: 10.1136/bmjopen-2024-093989. PMID 40721262
- [Derived] Pita TP, Misra S, Madonsela T, Tshazi A, Bosman S, Ayakaka I, Vlieghe E, Decroo T, Reither K, van Heerden A, Gils T. "If your CD4 count lowers, that is when you are similar to a person that is non-existent" A qualitative exploration of perceptions around advanced HIV disease in South Africa. BMC Public Health. 2025 Jul 3;25(1):2325. doi: 10.1186/s12889-025-23588-1. PMID 40610975
- See also: Project website — https://tbtriage.com/